CLINICAL TRIAL: NCT03443401
Title: Correlation of Trust and Outcomes Following Physical Therapy for Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of South Dakota (Other)
Collaborators: Iowa Physical Therapy Foundation (Other)
Responsible Party: Principal Investigator, Kory Zimney, PT, DPT, PhD, Assistant Professor, University of South Dakota
Other Study IDs: 2017.154
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Trust; Chronic Low Back Pain; Physical Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient participants: patients with chronic low back pain receiving standard physical therapy care
  Interventions: Procedure: Standard physical therapy care
- Physical Therapy clinician participants: Licensed physical therapist that is providing standard physical therapy care for a patient participant
  Interventions: Procedure: Standard physical therapy care

INTERVENTIONS:
Procedure: Standard physical therapy care — standard plan of care delivered to patient with chronic low back within scope of licensure

SUMMARY:
To investigate whether changes in trust between physical therapist and patient correlate to outcomes after receiving physical therapy care. We will be utilizing established questionnaires from the medical literature and one new generated questionnaire.

DETAILED DESCRIPTION:
1. The clinic site staff and physical therapist will fill out facility consent form to participate as a treatment site. The treating physical therapist participant will complete an informed consent form at their clinic site, if willing to participate via phone call with PI. If they consent, they will fill in a demographics form and be given an ID# that will be used for data collection by PI after informed consent received. This will take about 5 minutes.
2. Front office staff at each physical therapy clinic will provide recruitment letter for each new patient that potentially meets inclusion/exclusion criteria (coming into the clinic with low back that has persisted for greater than 3 month). If patient agrees to participate, they will fill out informed consent and HIPPA form on-line via PsychData link provided to them by clinic staff.
3. After completing the informed consent process, the patient participant will complete the necessary forms provided in PsychData link prior to the initial visit (Baseline demographics, General Trust in Physician Scale, Wake Forest Scale, Trust in Physician Scale, Patient Care Assessment Survey, Modified Oswestry Disability Index, Numeric Pain Rating Scale) Completing the forms will take place in the waiting room as they fill out their other normal initial paperwork needed for clinic site. This should take about 10-15 minutes. The forms will be handled electronically as the information is placed in the PI's individual PsychData account. The therapist participants will be blinded to research questionnaires information through the whole research project.
4. The patient then will receive a normal physical therapy initial evaluation and treatment as directed by the physical therapist based on the patient presentation.
5. At the conclusion of the initial visit, the patient participant will complete the necessary forms on-line through a second PsychData link (Wake Forest Scale, Trust in Physician Scale, Patient Care Assessment Survey, Working Alliance Inventory - Short Revised). This should take about 5-10 minutes.
6. Participant will continue to receive normal physical therapy care as directed by the physical therapist based on patient presentation. The majority of the visits (80%) have to be with the initial physical therapist involved in the care of the patient for that patient participant to be eligible for the study. The patient participant will still be eligible for all the gift cards even if they are eventually excluded due to not seeing the same therapist for 80% of the visits.
7. At the conclusion of care for the current episode (or at the end of 6 months of continual care by the provider), the patient participant will fill out forms on line to a third PsychData link (Wake Forest Scale, Trust in Physician Scale, Patient Care Assessment Survey, Working Alliance Inventory - Short Revised, Modified Oswestry Disability Index, Numeric Pain Rating Scale, Global Rate of Change). This should take about 10-15 minutes. If the patient is a no show and does not return for follow up visits, the principle investigator will send follow up letters to try to get final surveys completed.
8. After the second visit, the treating physical therapist will complete a PT Survey of Patient Connection and Engagement form on the patient via an on-line PyschData link. This will take less than 5 minutes. Treating therapist participant will be notified by PI that patient has consented into the study. This on-line PsychData information will be kept confidential from the patient participant.
9. At the conclusion of care (or 6 month time period), the physical therapist and clinic site will complete appropriate forms (PT Survey of Patient Connection and Engagement, number of visits, compliance (no show/cancellations), discharge disposition, and Current Procedural Terminology (CPT) billing codes for patients care) and send back to the principle investigator.

ELIGIBILITY:
Inclusion Criteria:

* age range 18 years of age or older, able to speak and read English, seeking physical therapy treatment for persistent low back pain of 3 months or greater. Being treated by a PT participant in the study

Exclusion Criteria:

* younger than 18 years of age, unable to speak or read English, patient needing to be referred out at any time for different level of medical care, concurrent pregnancy or cancer diagnosis, initial treating physical therapist does not see patient for 80% of treatments during episode of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients coming to seek care for chronic low back at outpatient physical therapy clinics
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kory J Zimney, DPT, Principal Investigator — University of South Dakota; Emilio J Puentedura, DPT, PhD, Study Chair — University of Nevada, Las Vegas; Morey Kolber, PT, PhD, Study Director — Nova Southeastern University; Adriaan Louw, PT, PhD, Study Director — International Spine and Pain Institute
Locations (11):
- United States (11):
  - One Accord Physical Therapy Casa Grande, Casa Grande, Arizona
  - Foothills Sports Medicine Physical Therapy, Phoenix, Arizona
  - Butte Premier Physical Therapy, Chico, California
  - Signature Physical Therapy, San Clemente, California
  - Rock Valley Physical Therapy, Silvis, Illinois
  - Hackensack Meridian Health-Mountainside Medical Center, Montclair, New Jersey
  - Miriam Hospital Outpatient Rehab, Providence, Rhode Island
  - PRO Physical Therapy, Winchester, Virginia
  - Outpatient Physical Therapy, Kent, Washington
  - Kitsap Physical Therapy and Sports Clinic, Silverdale, Washington
  - Phileo Health, Altoona, Wisconsin

IPD SHARING:
Plan to Share IPD: No
All data will be used as part of research project for dissertation purposes and not shared to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Participants
Started | 43
Completed | 29
Not Completed | 14
Not completed — Lost to Follow-up | 13
Not completed — Influential outlier | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Care Assessment Survey
Description: Measurement of trust of patient toward provider during clinical encounter. Minimum score of 8, maximal score of 40. Questions 1-7 are scored with a 5-point Likert scale, Question 8 is scored with a 11-point Likert scale. Higher score indicate better levels of trust.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 3.3 (1.1)

2. Primary Outcome: Change in Wake Forest Scale
Description: Measurement of trust of patient toward provider during clinical encounter. 10 item scale using a 5-point Likert scale. Score range from 10-50, with higher score indicating higher levels of trust.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 4.2 (1.5)

3. Primary Outcome: Change in Trust in Physician Scale
Description: Measurement of trust of patient toward provider during clinical encounter. 11 item scale using 5-point Likert scale. Score range from 11-55, with higher score indicating higher levels of trust.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 5.2 (.5)

4. Primary Outcome: Change in Oswestry Disability Index 2.0
Description: Measurement of function for individuals with low back pain. 10 categories with 6 statements scoring (0-5) for function. Raw scores range from 0-50, they are divided by highest possible score to produce a percentage. Lower percentage demonstrates less disability.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 11.1 (17.7)

5. Primary Outcome: Change in Numeric Pain Rating Scale
Description: Pain measurement scale. Measurement on 11-point scale from 0= no pain to 10= worst pain imaginable. Measure current, best in last 24 hours, and worst in last 24 hours and take average of all 3 measurements. Lower score represents lower pain rating.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 1.1 (2.6)

6. Primary Outcome: Global Rate of Change
Description: Global measurement of change of status during care. 11-point scale used (-5=very much worse, 0 = unchanged, 5 = completely recovered). Higher score represents better recovery.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 2.3 (.5)

7. Secondary Outcome: General Trust in Physician Scale
Description: global trust measurement of patient, 11 item scale using 5 point Likert scale. Minimum score 11, maximum score 55. Higher values, higher levels of trust. No subscales.
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 43.89 (6.27)

8. Secondary Outcome: Change in Working Alliance Inventory - Short Revised
Description: therapeutic alliance measurement. 12 item short form utilizing 5 point Likert scale. minimum score 12, maximum score 60. Higher score means higher therapeutic (working) alliance.
Time Frame: after initial visit and discontinuation of services, an average of 4-8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 5.6 (2.3)
Statistical Analysis 1: Comparison: Patient Participants; Test type: Superiority; p = 0.004, Spearman's rho — level of significance at <0.05; Mean Difference (Net) = 80

9. Secondary Outcome: Change in PT Survey of Patient Connection and Engagement
Description: Questionnaire completed by PT regarding their perceptions of the patients connection and engagement during the course of care. 10 question survey, using 5 point Likert scale. minimum score 10, maximum score 50. Higher score demonstrates higher patient connection and engagement.
Time Frame: after 2nd visit and discontinuation of services, an average of 4-8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 29
score on a scale | 0 (.5)
Statistical Analysis 1: Comparison: Patient Participants; Test type: Superiority; p = 0.027, Spearman's rho — Level of significance <0.05; Mean Difference (Net) = 80

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patient Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03443401/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03443401/ICF_001.pdf